CLINICAL TRIAL: NCT00418249
Title: Phase 2 Study of Topical AS101 for the Treatment of FAGA (Female Androgenetic Alopecia) in Menopause Women
Brief Title: Topical AS101 for Treatment of FAGA (Female Androgenetic Alopecia) in Menopause Women
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #69 REV 00
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2006-12

CONDITIONS: Alopecia
Keywords: Androgenetic Alopecia; Telogen effluvium; Chronic telogen effluvium; Menopause; Female Androgenetic Alopecia (FAGA)
MeSH Terms: conditions — Alopecia | interventions — ammonium trichloro(dioxoethylene-O,O'-)tellurate

INTERVENTIONS:
Drug: AS101

SUMMARY:
The primary objective of this study is to assess the safety and efficacy of topical AS101 as treatment for Female Androgenetic Alopecia (FAGA) in menopause women.

ELIGIBILITY:
Inclusion Criteria:

* Women in menopause, over 50 years of age.
* Clinically diagnosed for AGA, according to Ludwig scale I-II.

Exclusion Criteria:

* Women treated with chronic medications.
* Use of Minoxidil within 3 months prior to entering study.
* Women who have underwent hair transplantation.
* Use of drugs with androgenic or anti-androgenic effects.
* Any other type of hair loss.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40

PRIMARY OUTCOMES:
hair density

SECONDARY OUTCOMES:
Hair diameter, anagen/telogen ratio and hair growth rate,Global photographic assessment according to Female-Ludwig scale,
Self-administered satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Danny Ben-Amitai, M.D., Principal Investigator — Rabin Medical Center
Locations (1):
- Tel Aviv, Israel